CLINICAL TRIAL: NCT02374034
Title: Effect of Egoscue Corrective Exercise Prescription on Acute and Short-term Chronic Knee and Hip Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham Young University (Other)
Responsible Party: Principal Investigator, Ron Hager, Associate Professor, Brigham Young University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X13-0032
Record Dates: First submitted 2015-02-12; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Experimental group (n=20) completed a corrective exercise routine, as per the Egoscue Method, at least five days per week for two weeks.
  Interventions: Other: Corrective exercise
- Control (No Intervention): The control group maintained their current lifestyle for the two-week duration of the study.

INTERVENTIONS:
Other: Corrective exercise — Participants were assigned to either the exercise group, which performed Egoscue corrective exercises for two weeks, or the control group, which did not receive any treatment for two weeks.
  Arms: Treatment

SUMMARY:
The primary purpose of this experimental study was to determine the acute effect following one treatment and the short-term effect after a two-week program of Egoscue corrective exercises on chronic knee and hip pain.

DETAILED DESCRIPTION:
Participants for this study were recruited from the university community via email announcements and flyers. Participants were adults with chronic knee and/or hip pain. Chronic pain was defined as pain on most days of the week for at least 12 weeks. Individuals were excluded from the study if they (a) had undergone a knee or hip surgery or had sustained a knee or hip injury in the past 12 months, (b) were currently receiving any form of pain treatment such as physiotherapy, chiropractic, intraarticular injections, or prescription pain medications, (c) exhibited a severe lack of mobility, (d) reported an initial pain level < 3 cm on the Visual Analog Scale (VAS) scale, (e) were pregnant, or (f) were unable to understand English. Individuals were not excluded from participation if they were taking non-prescription drugs such as nonsteroidal anti-inflammatory drugs, although they were required to refrain from taking any pain medication during the 12 hours preceding the first, and subsequent assessments. A power analysis using a power level of 80% and alpha set at 0.05 indicated a sample size of 40 participants (20 in the control group and 20 in the exercise group). A large effect size (0.80) was assumed because this has been reported in the literature26 for differences in Western Ontario and McMaster Universities Arthritis Index (WOMAC) scores following an at-home exercise program. Forty-two eligible participants were originally recruited.

All participants completed a pre-participation questionnaire that included questions about age, gender, injuries, pain medication use, and previous or planned total hip and/or knee arthroplasty. Participants completed two versions of the VAS for knee and/or hip pain: one for pain at rest and one for pain during movement. If participants had pain in multiple joints, they were told to record their overall level of pain. Participants were told to indicate their "usual pain" over the past seven days. Participants needed to have a VAS pain score of at least 3 cm (either at rest or during movement) in order to participate in the study. Participants also completed the WOMAC at the time of the visit. Participants' body mass was measured to the nearest 0.1 kg and height to the nearest 0.5 cm using a digital scale and a stadiometer, respectively.

Egoscue Method protocol was followed and a postural alignment specialist trained in postural evaluation conducted an assessment. To reduce possible inter-rater error, the same researcher conducted all postural evaluations. An individualized exercise program (E-cise menu) was generated using the ePeteTM software (version 4.4.3) based on the noted postural deviations. To ensure that all participants were prescribed the same volume of exercise, the E-cise menus were adjusted by adding or removing exercises so the time required to complete the exercises was approximately 45 minutes.

Participants in the exercise group were led through their complete E-cise menu by the researcher to ensure competency on the exercises. Participants in the control group did not perform any exercises for 45 minutes. Following the first exercise session or 45 minutes of rest, participants completed the VAS again for their current knee and/or hip pain at rest and with movement.

All participants were given logs (one for each day of the week), which they were to fill out every evening before retiring to bed. These logs contained questions about their compliance to the E-cise menu (for those in the exercise group), pain medication use, and a VAS for pain at rest and during movement. Participants in the control group were instructed to maintain their current lifestyle for the two week duration of the study and a return visit was scheduled one week later. Participants in the exercise group were scheduled for a return visit the following day so that E-cises could be observed for competency and any adjustments could be made to the E-cise menu if participants were experiencing pain during an E-cise. Participants in the exercise group were instructed to complete their E-cise menu at home on at least five days of the week, but preferably every day, for the next two weeks.

All participants were assessed and evaluated on all variables previously mentioned at the end of week number 1 and again at the end of the study after week number 2. Participants in the control group were given a personalized E-cise menu, along with instructions, at this time.

ELIGIBILITY:
Inclusion Criteria:

* participants with either or both of chronic hip and knee pain
* pain will be defined as pain on most days of the week for at least 12 weeks

Exclusion Criteria:

* undergone a knee or hip surgery or had sustained a knee or hip injury in the past 12 months
* currently receiving any form of pain treatment such as physiotherapy, chiropractic, intraarticular injections, or prescription pain medications
* exhibited a severe lack of mobility
* reported an initial pain level < 3 cm on the Visual Analog Scale (VAS) scale
* pregnant
* unable to understand English

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in function and pain | two weeks
  Pain and function will be assessed with the WOMAC, a self-administered, multidimensional questionnaire

SECONDARY OUTCOMES:
Changes in daily pain | two weeks
  The VAS will be daily to assess changes in pain over a two week period

REFERENCES:
- [Background] Hootman JM, Helmick CG. Projections of US prevalence of arthritis and associated activity limitations. Arthritis Rheum. 2006 Jan;54(1):226-9. doi: 10.1002/art.21562. PMID 16385518
- [Background] Verhaak PFM, Kerssens JJ, Dekker J, Sorbi MJ, Bensing JM. Prevalence of chronic benign pain disorder among adults: a review of the literature. Pain. 1998 Sep;77(3):231-239. doi: 10.1016/S0304-3959(98)00117-1. PMID 9808348
- [Background] Griegel-Morris P, Larson K, Mueller-Klaus K, Oatis CA. Incidence of common postural abnormalities in the cervical, shoulder, and thoracic regions and their association with pain in two age groups of healthy subjects. Phys Ther. 1992 Jun;72(6):425-31. doi: 10.1093/ptj/72.6.425. PMID 1589462
- [Background] Kuo YL, Tully EA, Galea MP. Sagittal spinal posture after Pilates-based exercise in healthy older adults. Spine (Phila Pa 1976). 2009 May 1;34(10):1046-51. doi: 10.1097/BRS.0b013e31819c11f8. PMID 19404180
- [Background] Hernandez-Molina G, Reichenbach S, Zhang B, Lavalley M, Felson DT. Effect of therapeutic exercise for hip osteoarthritis pain: results of a meta-analysis. Arthritis Rheum. 2008 Sep 15;59(9):1221-8. doi: 10.1002/art.24010. PMID 18759315
- [Background] Ferraz MB, Quaresma MR, Aquino LR, Atra E, Tugwell P, Goldsmith CH. Reliability of pain scales in the assessment of literate and illiterate patients with rheumatoid arthritis. J Rheumatol. 1990 Aug;17(8):1022-4. PMID 2213777